CLINICAL TRIAL: NCT06114758
Title: The Comparison of the Effectiveness of Rectal Misoprostol and Intravenous Tranexamic Acid in Reducing Intraoperative Bleeding in Patients Undergoing Myomectomy
Brief Title: Comparison Effectiveness of Rectal Misoprostol & Intravenous Tranexamic Acid Reducing Hemorrhage in Myomectomy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Tuğba Ağbal, clinical doctor, Ankara Etlik City Hospital
Other Study IDs: AEŞH-EK1-2023-383
Record Dates: First submitted 2023-10-18; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Hemorrhage, Surgical; Myoma;Uterus; Effect of Drug; Postoperative Hemorrhage; Postoperative Complications
Keywords: myoma uteri; fibroids; hemmorhage; prostoglandinf2α; tranexamic acid
MeSH Terms: conditions — Blood Loss, Surgical; Myofibroma; Postoperative Hemorrhage; Postoperative Complications; Leiomyoma | interventions — Misoprostol; Tablets; Tranylcypromine; Tranexamic Acid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- control group - group 1: 1. Patients' postoperative 1st, 2nd, and 6th-hour vital signs (pulse rate, systolic and diastolic blood pressure, temperature, oxygen saturation).
  2. Shock indices.
  3. Hemogram and hematocrit values at 6-24 hours postoperatively.
  4. Duration of the surgery.
  5. Adverse effects experienced by the patients.
  6. Additional treatments administered.
  7. Whether blood transfusion was performed or not.
- intraoperatively admistiration of tranexamic acid (1 gram intravenous) - group 2: 1. Patients' postoperative 1st, 2nd, and 6th-hour vital signs (pulse rate, systolic and diastolic blood pressure, temperature, oxygen saturation).
  2. Shock indices.
  3. Hemogram and hematocrit values at 6-24 hours postoperatively.
  4. Duration of the surgery.
  5. Adverse effects experienced by the patients.
  6. Additional treatments administered.
  7. Whether blood transfusion was performed or not.
  Interventions: Drug: Transamine
- intraoperatively admistiration of prostoglandin f2 alfa (cytotec 400 microgram rectal)- group 2: 1. Patients' postoperative 1st, 2nd, and 6th-hour vital signs (pulse rate, systolic and diastolic blood pressure, temperature, oxygen saturation).
  2. Shock indices.
  3. Hemogram and hematocrit values at 6-24 hours postoperatively.
  4. Duration of the surgery.
  5. Adverse effects experienced by the patients.
  6. Additional treatments administered.
  7. Whether blood transfusion was performed or not.
  Interventions: Drug: Cytotec 200Mcg Tablet

INTERVENTIONS:
Drug: Cytotec 200Mcg Tablet — the admistiration of 400 Mcg rectal cytotec while starting the surgery, just before the patient is covered
  Other Names: misoprostol; prostoglandin f2α
  Groups: intraoperatively admistiration of prostoglandin f2 alfa (cytotec 400 microgram rectal)- group 2
Drug: Transamine — 1 gram intravenous slow infusion intraoperatively as we start the laparatomy
  Other Names: tranexamic acid
  Groups: intraoperatively admistiration of tranexamic acid (1 gram intravenous) - group 2

SUMMARY:
Fibroids are the most commonly encountered tumors in the female reproductive system. In patients, fibroids most often lead to abnormal uterine bleeding and the resulting anemia. In some cases, they can cause infertility or habitual abortions. Another complaint caused by fibroids is pain due to pressure and effects on adjacent organs. Very large fibroids can lead to abdominal swelling. Therefore, if a patient becomes symptomatic due to fibroids, myomectomy or, if necessary, hysterectomy is required.

Because fibroids have a significant blood supply, there is a high risk of intraoperative bleeding and related complications. Additionally, the most common complication in these patients after the operation is bleeding. In many of these patients, intraoperative or postoperative blood transfusions are performed. If bleeding cannot be intervened early in these patients, hemodynamic instability, shock, coagulopathy, and, in the final stage, death can occur due to hemorrhage. Therefore, both intraoperative and postoperative bleeding control is of vital importance in patients undergoing myomectomy.

DETAILED DESCRIPTION:
In this study, data of patients admitted with a diagnosis of uterine fibroids to the Department of Obstetrics and Gynecology, Women's Health and Obstetrics (EŞH) between September 1, 2022, and Sempember 1, 2024, who underwent myomectomy (either laparotomic or laparoscopic), will be collected.

The parameters to be examined in the research are as follows:

1. Patients' postoperative 1st, 2nd, and 6th-hour vital signs (pulse rate, systolic and diastolic blood pressure, temperature, oxygen saturation).
2. Shock indices.
3. Hemogram and hematocrit values at 6-24 hours postoperatively.
4. Duration of the surgery.
5. Adverse effects experienced by the patients.
6. Additional treatments administered.
7. Whether blood transfusion was performed or not.

In this study, the G-power analysis program was used to determine the minimum sample size, taking into account a 10% margin of error. According to the analysis results, the minimum number of patients to be included in the study for a total of 75 patients across 3 groups was determined. Statistical analysis of the data obtained in the study will be conducted using the SPSS Statistics 22 software package. A 95% confidence interval will be calculated for each variable, and results will be considered statistically significant for p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Laparotomic myomectomy surgeries
* Laparoscopic myomectomy surgeries

Exclusion Criteria:

* Identifying missing or suspicious data related to the patient
* Administering both intraoperative and postoperative medications to the patient

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women
Study Population: In our study, data of patients admitted with a diagnosis of uterine fibroids to the Department of Obstetrics and Gynecology, Women's Health and Obstetrics (Etlik City Hospital) between October 1, 2023, and October 1, 2024, who underwent myomectomy (either laparotomic or laparoscopic), will be collected prospectively
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of patients' preoperative and postoperative hemogram levels | 24 hours
  The basal hemogram levels ( gr/dL) of the patients will be compared with the hemogram levels at 6 and 24 hours.
Comparison of patients' preoperative and postoperative hematocrit levels | 24 hours
  The basal hematocrit levels (%) of the patients will be compared with the hematocrit levels at 6 and 24 hours.
Comparison of patients' postoperative shock indices | 6 hour
  postoperative 1st, 2nd, and 6th-hour shock indices (heart rate (beats in minute) / systolic blood pressure(mmHg) ) will be compared

SECONDARY OUTCOMES:
Comparison of the patients' postoperative heart rate | 6 hour
  Patients postoperative 1st, 2nd, and 6th-hour heart rate (beats in minute) will be compared
Comparison of the patients' postoperative systolic and diastolic blood pressure | 6 hour
  Patients postoperative 1st, 2nd, and 6th-hour systolic and diastolic blood pressure (mmHg) will be compared

CONTACTS AND LOCATIONS:
Locations (1):
- Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No